CLINICAL TRIAL: NCT04097119
Title: Impact of a Dietary Supplement to Support HDL Function on Safety Markers and Quality of Life
Brief Title: HDL Function Dietary Supplement Safety and QOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Metagenics, Inc. (Industry)
Collaborators: Hypertension Institute, Nashville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-035-HDL
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: HDL; Health, Subjective
Keywords: HDL function; HDL dysfunction; nutritional supplement; quality of life; dietary supplement
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary supplement arm (Other): Subjects to receive a specific dietary supplement
  Interventions: Dietary Supplement: Dietary supplementation

INTERVENTIONS:
Dietary Supplement: Dietary supplementation — Subjects receive a specific dietary supplementation designed to support HDL function daily for 12 weeks

SUMMARY:
Nutritional supplements are routinely purchased by consumers with suboptimal HDL to support their health, lifestyle and overall quality of life. Many such products receive minimal evaluation prior to marketing. This study aims to evaluate a specific nutritional supplement for its safety, tolerance and acceptability as well as the potential for positive impact on quality of life.

DETAILED DESCRIPTION:
High density lipoprotein cholesterol (HDL), often considered the 'good cholesterol,' plays an essential role in reverse cholesterol transport (RCT), and has anti-inflammatory, anti-oxidative, and anti-thrombotic actions in the body. However, studies have shown that higher HDL cholesterol (HDL-C) levels are not always cardioprotective, and that the functionality of the HDL molecule is critical for cardioprotection.

The HDL molecule is associated with many proteins (the HDL proteome) such as apolipoprotein A-one (apoA-I) and paraoxonase (PON) which are critical for its function. These proteins can be the target of oxidative damage which negatively impacts HDL functionality. Loss of HDL function leads to impaired RCT and the build of cholesterol within the vasculature with an increased risk of atherosclerotic plaque development. Gain of HDL dysfunction leads to HDL acting as a pro-inflammatory and pro-oxidant molecule, further increasing cardiovascular risk.

Several dietary ingredients have been shown to support various aspects of HDL function and the HDL proteome. Examples include pomegranate juice and extract, lycopene, and quercetin.

Nutritional supplements are routinely purchased by consumers with suboptimal HDL to support their health, lifestyle and overall quality of life. Many such products receive minimal evaluation prior to marketing. As part of the investigator's commitment to safe and beneficial formulating of nutritional supplements, an evaluation of both the safety, tolerance and acceptability as well as the potential for positive impact on quality of life, this study aims to collect information on relevant outcomes related to quality of life and recovery, with a view to understanding potential for benefit and areas for larger research focus.

ELIGIBILITY:
Inclusion Criteria:

* Men: Total HDL of equal to or less than 38 mg / dL in men AND a low HDL-P of less than or equal to 7200 by Spectracell LPP Plus.
* Women: Total HDL equal to or less than 45 mg/dl in women, AND a low HDL-P of less than or equal to 7200 by Spectracell LPP Plus.
* Willingness to maintain current lifestyle (diet and exercise) practices
* Willingness to eat fish no more than twice per week and keep intake stable throughout the study
* Willingness to give written informed consent to participate in the study
* Willingness to follow lifestyle instructions for 24 hours prior to the study visit.
* No known food allergy or intolerance to the ingredients in the study product (fish, shellfish)
* Not currently taking (washout of at least 30 days required) any other supplements that would interfere with the study results
* Not currently taking (washout of at least 30 days required) any other supplements designed to support HDL.

Exclusion Criteria:

* Use of medications classified as narcotics 30 days prior to Screening and for the duration of the study.
* Use of an investigational drug or participation in an investigational study within 30 days prior to Day 1 and for the duration of the study.
* Current use (at least 30 days wash-out required) of any lipid lowering medication which, in the view of the PI, may interfere with the results.
* Known allergy or hypersensitivity to study product.
* No initiation of a new or change of an existing exercise regimen within 15 days prior to Day 1 and for the duration of the study.
* No initiation of a new or change of an existing food plan 30 days prior to Day 1 and for the duration of the study.
* No current involvement or within 30 days of Day 1 of a significant diet or weight loss program such as Atkin's or other Low-Carb diet programs, very low calorie liquid diet programs (such as Optifast, Medifast and/or HMR) or any diet that has led to a weight loss of 5% of body weight over a period of 10 weeks.
* No serious, unstable illnesses including cardiovascular, hepatic, renal, gastrointestinal, respiratory, endocrine, neurologic, immunologic, or hematologic disease.
* Known infection with Human Immunodeficiency Virus (HIV), Tuberculosis or Hepatitis B or C.
* Subjects with a current diagnosis or personal history of:

  * Previous myocardial infarction within 5 years, Unstable angina, Previous stroke or transient ischemic attack (TIA) within 5 years, Uncompensated congestive heart failure, Previous percutaneous transluminal coronary angioplasty (PCTA) or stent within 5 years, Previous coronary artery bypass grafts (CABG) within 5 years
  * Type 1 diabetes mellitus
  * Any significant liver or kidney disease such as cirrhosis or non-alcoholic fatty liver disease, glomerulonephritis, and/or undergoing dialysis treatment. Cr over 2.5 mg/dL.
  * Any malignancy (with the exception of basal or squamous cell carcinoma of the skin if adequately treated and no recurrence for >5 years).
  * Any serious mental illness including depression, manic episodes, post-traumatic disorder, obsessive-compulsive disorder, personality disorders, history of attempted suicide or violence within 12 months prior to Screening and for the duration of the study.
  * Any personal history of bipolar disorders, schizophrenia or psychotic behaviors.
  * Personal history of seizure disorder other than a single childhood febrile seizure that fully resolved.
  * Known presence of raised intraocular pressure or history of narrow angle glaucoma.
  * A major medical or surgical event requiring hospitalization within the preceding 3 months
  * The presence of any disease which influences digestion and absorption of nutrients
  * History of any bariatric surgery procedure
* Consumption of alcohol the evening prior to any study visit
* Use of drugs of abuse (such as marijuana, cocaine, phencyclidine [PCP] and methamphetamine) within 12 months prior to Screening and for the duration of the study.
* History of alcohol abuse or a diagnosis of alcoholism within 12 months prior to Screening and for the duration of the study.
* Inability to comply with study and/or follow-up visits.
* Any other concurrent condition which, in the opinion of the Investigator, would preclude participation in this study or interfere with compliance.
* Pregnancy
* Females of child bearing age not on an accepted contraception control method

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of participant adverse events during the supplementation period | 0 - week 12
  Tolerability of oral intake of the supplement will primarily be evaluated by determining the frequency of adverse events during the supplementation period

SECONDARY OUTCOMES:
Medical Outcomes Study Short Form 36 (MOS SF-36) questionnaire | 0 - week 12
  The MOS SF-36 is an indicator of overall health status. It has an eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability.
Patient-Reported Outcomes Measurement Information System (PROMIS-43) questionnaire | 0 - week 12
  Patient-Reported Outcomes Measurement Information System (PROMIS-43) is a qualitative measure of an individual's quality of life. The questions are categorized into seven domains (Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities). A T-score in each domain will be generated based on individual's answer. A score of 50 with standard deviation of 10 reflects the general population, from which the individual's score will be compared to determine improvement or lack of.
Rate of HDL function | 0 - week 12
  A blood test developed by Cleveland Heart Lab that reflects the function of HDL particle
Profile (amount) of HDL map | 0 - week 12
  A blood test developed by Boston Heart Diagnostics that quantifies the amount of apoA-I in the five most significant HDL subpopulations, resulting in a deeper understanding of a patient's cardiovascular disease risk.
Concentration of hsCRP | 0 - week 12
  A blood test that measures high-sensitivity C-reactive protein (hsCRP)
Concentration of MPO | 0 - week 12
  A blood test that measures myeloperoxidase (MPO)
Concentration of HDL-C | 0 - week 12
  A blood test that measures high-density lipoprotein cholesterol (HDL-C) level
Number of HDL-P | 0 - week 12
  A blood test that measures high-density lipoprotein cholesterol (HDL-C) particle number

CONTACTS AND LOCATIONS:
Overall Officials: Mark Houston, MD, Principal Investigator — Hypertension Institute
Locations (1):
- Hypertension Institute, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No